CLINICAL TRIAL: NCT04432922
Title: Perceptions, Representations and Experiences of Septic Isolation of Hospitalized
Brief Title: Perceptions, Representations and Experiences of Septic Isolation of Hospitalized Patients for COVID-19 Infection
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Responsible Party: Sponsor
Other Study IDs: ISOCOV
Record Dates: First submitted 2020-06-15; First posted 2020-06-16 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: COVID19
Keywords: Septic isolation, perception, questionnaire
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Hospitalized Patients for COVID-19 Infection — Face to face semi-directed interviews about perceptions, representations and experiences of septic isolation, including nine opened-questions.

SUMMARY:
The aim of this study is to analyze the perceptions, representations and experiences of septic isolation of patients hospitalized for COVID-19 infection.

This analysis could lead to better understanding and communication between the medical profession and patients in septic isolation in hospital. It would also provide patient-specific responses to their expectations, as to their families.

DETAILED DESCRIPTION:
SARS-Cov2 is a new virus responsible for the COVID-19 pandemic. For the first time, it was observed in Wuhan, China in December 2019. For this previously unknown contagious disease, which can cause severe respiratory infections, isolation precautions in hospitals and public places are one of the cornerstones for fighting this pandemic.

Hospital isolation precautions have been present since the 19th century as a means to control the spread of infections. Septic isolation includes contact isolation, droplets and air. Isolation precautions must be prescribed by a physician. To our knowledge, there are few studies about the impact of septic isolation on hospitalized patients at both the psychological level and the relationship with doctors.

This study could enable a better understanding and communication between the medical profession and patients in septic isolation during hospitalization. It could also provide patient-specific responses to their expectations.

ELIGIBILITY:
Inclusion Criteria:

* Major patients
* Living in metropolitan France during the SARS-CoV2 pandemic
* Being or having been hospitalized in isolation contact and droplet for a COVID-19 infection (proven or suspected)
* Being in the process of leaving hospital
* Ready for No Opposition for Participation in the Protocol

Exclusion Criteria:

* Patients under guardianship or curatorship
* Patients unable to give free and informed consent;
* Patients under safeguarding justice
* Hospitalized patients on oxygen therapy with speech dyspnea

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be provided to Covid 19 participants during their hospitalization or upon discharge from hospitalization
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2020-11-15 (Actual); Study Completion 2020-11-15 (Actual)

PRIMARY OUTCOMES:
To highlight the perceptions, representations and experiences of septic isolation of patients hospitalized for COVID-19 infection | 1 day

SECONDARY OUTCOMES:
to identify key elements to improve the medical discourse on septic isolation among patients | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Centre hospitalier intercommunal de Villeneuve St Georges, Villeneuve-Saint-Georges, France

IPD SHARING:
Plan to Share IPD: No